CLINICAL TRIAL: NCT06917937
Title: Is Exercise Program Added to Corticosteroid Injection Effective on Pain and Performance in Plantar Fasciitis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Sevtap Cakir, Asst. Prof., Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSBU-PF
Record Dates: First submitted 2025-03-28; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Plantar Fascitis
Keywords: Foot; Foot Disease; Plantar Fasciitis; Exercise; Steroid
MeSH Terms: conditions — Foot Diseases; Fasciitis, Plantar; Motor Activity | interventions — Resistance Training; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: A prospective single-center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Exercise program in added on to corticosteroid injection (Group I) (Experimental): Our exercise program in our study; (i) foot intrinsic muscle strengthening exercise (with a load of 3 kg), (ii) plantar fascia stretching with finger extension, (iii) standing gastrocnemius muscle stretching, (iv) sitting achilles tendon stretching, (v) plantar fascia and gastrocnemius stretch on the step, (vi) cold massage exercise in the arch of the foot. We stated that the group to which exercise was added should do the exercises regularly for 6 weeks, in the specified number and time.
  Interventions: Other: Exercise Program; Other: Corticosteroid injection
- Corticosteroid injection (Group II) (Active Comparator): The orthopedic physician administered the corticosteroid injection as a mixture of 1 ml of arthropane (5 mg of triamcinolone hexacetonide) and 4 ml of citanest. Before the application, the physician cleaned the area to be treated with 10% povidone iodine. He made a single dose injection by entering the painful point determined by palpation around the calcaneal spur and plantar fascia from the percutaneous foot-heel lateral. The patients were in the prone position with the ankle in a neutral position.
  Interventions: Other: Corticosteroid injection

INTERVENTIONS:
Other: Exercise Program — Our exercise program in our study; (i) foot intrinsic muscle strengthening exercise (with a load of 3 kg), (ii) plantar fascia stretching with finger extension, (iii) standing gastrocnemius muscle stretching, (iv) sitting achilles tendon stretching, (v) plantar fascia and gastrocnemius stretch on the step, (vi) cold massage exercise in the arch of the foot. We stated that the group to which exercise was added should do the exercises regularly for 6 weeks, in the specified number and time.
  Arms: (Exercise program in added on to corticosteroid injection (Group I)
Other: Corticosteroid injection — The orthopedic physician administered the corticosteroid injection as a mixture of 1 ml of arthropane (5 mg of triamcinolone hexacetonide) and 4 ml of citanest. Before the application, the physician cleaned the area to be treated with 10% povidone iodine. He made a single dose injection by entering the painful point determined by palpation around the calcaneal spur and plantar fascia from the percutaneous foot-heel lateral. The patients were in the prone position with the ankle in a neutral position.
  After the application, he covered the area with a sterile cloth and said to remove it after 3 hours. He stated that patients could apply ice to the injected area if necessary for pain control, and advised patients to avoid all jogging and other high-impact activities on the day of injection. No additional treatments, including NSAIDs, orthoses, and night splints, were allowed during the study period.

SUMMARY:
Plantar fasciitis (PF) involves the degeneration of the medial calcaneal tuberosity and nearby perifascial tissues in the heel. It is the leading cause of heel pain, typically resulting from repetitive strain on the plantar fascia, causing structural damage. Key risk factors for PF include an increased body mass index in active individuals and a greater range of plantar flexion motion. Treatment options for PF vary, and there is no clear consensus on the most effective approach. Conservative treatments may include rest, stretching exercises for the plantar fascia and Achilles tendon, strengthening exercises for foot intrinsic muscles, nonsteroidal anti-inflammatory drugs (NSAIDs), orthotics, heel pads, dorsiflexion night splints, and corticosteroid injections. These treatments may be used individually or in combination. Corticosteroid injections are the most frequently used invasive treatment. However, there has been limited research examining the effects of corticosteroid injections combined with exercises targeting intrinsic foot muscle strength on functionality and walking distance. The objective of this study was to evaluate the impact of an exercise program added to corticosteroid injections on pain relief and functional performance in individuals with PF.

ELIGIBILITY:
Inclusion Criteria:

* Those over the age of 18
* Those who have pain in the plantar region for 1 month and this pain is 5 or more according to VAS,
* Those who describe pain on the first step of the morning,
* Those with plantar fascia tenderness on palpation,
* Patients who will be in harmony with the physician and physiotherapist in exercise and follow-up throughout the entire study period.

Exclusion Criteria:

* Cases with fracture, entrapment neuropathy and rupture,
* Those with neurological and systemic diseases,
* Those with a Body Mass Index (BMI) of more than 40,
* Conditions with a local contraindication to corticosteroid,
* Participants who have situations that may prevent their safety, execution or interpretation of the results during the continuation of the training and applied of the test protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-16 (Actual); Primary Completion 2019-03-03 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Muscle Shortness Tests | a day before the rehabilitation
  Plantar and Dorsi Flexion Flexibility, Gastrocnemius Shortness, Hamstring Shortness, Hip Flexor Shortness, Tensor Fascia Lata Shortness shortness tests were performed.
Muscle Shortness Tests | up to 3 weeks
  Plantar and Dorsi Flexion Flexibility, Gastrocnemius Shortness, Hamstring Shortness, Hip Flexor Shortness, Tensor Fascia Lata Shortness shortness tests were performed.
Muscle Shortness Tests | up to 6 weeks
  Plantar and Dorsi Flexion Flexibility, Gastrocnemius Shortness, Hamstring Shortness, Hip Flexor Shortness, Tensor Fascia Lata Shortness shortness tests were performed.
American Orthopedic Foot and Ankle Society Hindfoot Clinical Evaluation System (AOFAS- hindfoot) | a day before the rehabilitation
  The AOFAS hindfoot clinical assessment system evaluates the ankle, subtalar, talonavicular, and calcaneocuboid joints. The scoring system allocates 50 points for function, 40 points for pain, and 10 points for alignment. A higher score indicates a better condition for the patient.
American Orthopedic Foot and Ankle Society Hindfoot Clinical Evaluation System (AOFAS- hindfoot) | up to 3 weeks
  The AOFAS hindfoot clinical assessment system evaluates the ankle, subtalar, talonavicular, and calcaneocuboid joints. The scoring system allocates 50 points for function, 40 points for pain, and 10 points for alignment. A higher score indicates a better condition for the patient.
American Orthopedic Foot and Ankle Society Hindfoot Clinical Evaluation System (AOFAS- hindfoot) | up to 6 weeks
  The AOFAS hindfoot clinical assessment system evaluates the ankle, subtalar, talonavicular, and calcaneocuboid joints. The scoring system allocates 50 points for function, 40 points for pain, and 10 points for alignment. A higher score indicates a better condition for the patient.
American Orthopedic Foot and Ankle Society Midfoot Clinical Evaluation System (AOFAS- midfoot) | a day before the rehabilitation
  This scale allocates 45 points for function, 40 points for pain, and 15 points for alignment. Higher scores indicate that the patient's condition is favorable.
American Orthopedic Foot and Ankle Society Midfoot Clinical Evaluation System (AOFAS- midfoot) | up to 3 weeks
  This scale allocates 45 points for function, 40 points for pain, and 15 points for alignment. Higher scores indicate that the patient's condition is favorable.
American Orthopedic Foot and Ankle Society Midfoot Clinical Evaluation System (AOFAS- midfoot) | up to 6 weeks
  This scale allocates 45 points for function, 40 points for pain, and 15 points for alignment. Higher scores indicate that the patient's condition is favorable.
Foot Function Index | a day before the rehabilitation
  It is a 23-item questionnaire designed to assess how foot pathology affects pain, disability, and activity limitations. The FFI score was calculated based on 5 questions related to pain (with a maximum of 50 points). Each question was scored on a scale from 0 to 10, where 0 represents no pain and 10 indicates unbearable pain. In our study, we utilized the Turkish version of the FFI questionnaire.
Foot Function Index | up to 3 weeks
  It is a 23-item questionnaire designed to assess how foot pathology affects pain, disability, and activity limitations. The FFI score was calculated based on 5 questions related to pain (with a maximum of 50 points). Each question was scored on a scale from 0 to 10, where 0 represents no pain and 10 indicates unbearable pain. In our study, we utilized the Turkish version of the FFI questionnaire.
Foot Function Index | up to 6 weeks
  It is a 23-item questionnaire designed to assess how foot pathology affects pain, disability, and activity limitations. The FFI score was calculated based on 5 questions related to pain (with a maximum of 50 points). Each question was scored on a scale from 0 to 10, where 0 represents no pain and 10 indicates unbearable pain. In our study, we utilized the Turkish version of the FFI questionnaire.
6-minute walk test | a day before the rehabilitation
  The 6MWT is a simple, safe, and well-tolerated test that effectively reflects daily life activities. In our study, the 6MWT was conducted in a 30-meter long, flat, enclosed corridor. We measured the patient's heart rate, respiratory rate, and blood pressure before the test, immediately after completion, and again 5 minutes later. Fatigue levels were evaluated using the Borg Scale, and the distance walked by the patient was recorded in meters.
6-minute walk test | up to 3 weeks
  The 6MWT is a simple, safe, and well-tolerated test that effectively reflects daily life activities. In our study, the 6MWT was conducted in a 30-meter long, flat, enclosed corridor. We measured the patient's heart rate, respiratory rate, and blood pressure before the test, immediately after completion, and again 5 minutes later. Fatigue levels were evaluated using the Borg Scale, and the distance walked by the patient was recorded in meters.
6-minute walk test | up to 6 weeks
  The 6MWT is a simple, safe, and well-tolerated test that effectively reflects daily life activities. In our study, the 6MWT was conducted in a 30-meter long, flat, enclosed corridor. We measured the patient's heart rate, respiratory rate, and blood pressure before the test, immediately after completion, and again 5 minutes later. Fatigue levels were evaluated using the Borg Scale, and the distance walked by the patient was recorded in meters.
50 meters walking test | a day before the rehabilitation
  The test evaluates walking ability, and patients were instructed to walk at their own comfortable pace for a distance of 50 meters. The stopwatch was started with the command to begin at the starting point. Upon reaching the 50-meter mark, we stopped the stopwatch and recorded the time.
50 meters walking test | up to 3 weeks
  The test evaluates walking ability, and patients were instructed to walk at their own comfortable pace for a distance of 50 meters. The stopwatch was started with the command to begin at the starting point. Upon reaching the 50-meter mark, we stopped the stopwatch and recorded the time.
50 meters walking test | up to 6 weeks
  The test evaluates walking ability, and patients were instructed to walk at their own comfortable pace for a distance of 50 meters. The stopwatch was started with the command to begin at the starting point. Upon reaching the 50-meter mark, we stopped the stopwatch and recorded the time.
Visual Analogue Scale | a day before the rehabilitation
  Patients were asked to indicate their current pain level on a visual analog scale, which consisted of a 10 cm line. The distance was then measured using a ruler and recorded. A lower score indicates decreased pain.
Visual Analogue Scale | up to 3 weeks
  Patients were asked to indicate their current pain level on a visual analog scale, which consisted of a 10 cm line. The distance was then measured using a ruler and recorded. A lower score indicates decreased pain.
Visual Analogue Scale | up to 6 weeks
  Patients were asked to indicate their current pain level on a visual analog scale, which consisted of a 10 cm line. The distance was then measured using a ruler and recorded. A lower score indicates decreased pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No